CLINICAL TRIAL: NCT03432312
Title: A Single-Center, Single-Dose, Open-Label, Laboratory-Blind, Randomized, Two-Period Crossover Study to Determine the Bioequivalence of Two Nicotine Resinate Lozenge Formulations Containing Nicotine 4 mg in up to 42 Healthy Male and Female Smokers Under Fasting Conditions
Brief Title: Single-Dose Bioequivalence Study Comparing Two 4 mg Nicotine Lozenges
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fertin Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: F-ZA114
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine 4 mg mint lozenges (Experimental)
  Interventions: Drug: Nicotine lozenge
- NiQuitin 4 mg mint lozenges (Active Comparator)
  Interventions: Drug: Nicotine lozenge

INTERVENTIONS:
Drug: Nicotine lozenge — Nicotine mint lozenge, 4 mg
  Arms: Nicotine 4 mg mint lozenges
Drug: Nicotine lozenge — NiQuitin mint lozenge, 4 mg
  Arms: NiQuitin 4 mg mint lozenges

SUMMARY:
The purpose of the study is to compare the pharmacokinetic (PK) profiles and assess bioequivalence between a new nicotine lozenge and a reference nicotine lozenge in healthy smokers

ELIGIBILITY:
Inclusion Criteria:

1. Written consent given for participation in the study.
2. Healthy males and females, 18 to 55 years (inclusive) at screening.
3. Body Mass Index (BMI) between 18.5 and 30 kg/m2 (both inclusive).
4. Body mass not less than 50 kg.
5. Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
6. Females, if:

   * Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal, Note: in postmenopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.
   * Of childbearing potential, the following conditions are to be met:

   Negative pregnancy test

   If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received IMP, every attempt must be made to follow her to term.

   Not lactating

   Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study

   Examples of reliable methods of contraception include oral (documented that the dose has been stable for at least one month before the first intake of IMP), injectable or implantable contraceptives and non-hormonal intrauterine device.

   In this study the concomitant use of hormonal contraceptives is allowed. Other methods, if considered by the investigator as reliable, will be accepted.
7. History of cigarette smoking of at least 10 cigarettes per day continuously for the past 3 months prior to screening and smokes first cigarette in less than 30 minutes after waking up in the morning.
8. No use of any tobacco or nicotine-containing products within 21 days of the first dose except cigarettes.
9. Have no interest in quitting smoking.
10. Have accepted to refrain from smoking for the duration of the study periods.
11. Exhaled CO concentration > 10 ppm at screening.
12. Successfully completed the dissolution training session prior to randomization.
13. Ability to communicate and comply with all study requirements including the study specific method of administration for the nicotine lozenges.

Exclusion Criteria:

1. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
2. Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any IMP substance.
3. Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females or evidence of excessive alcohol use as indicated by an alcohol breathalyzer test result ≥ 0.01%.
4. Regular exposure to substances of abuse (other than alcohol) within the past year.
5. Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator.

   In this study the concomitant use of hormonal contraceptives is allowed.
6. Expired CO levels greater than 10 ppm in the morning prior to dosing.
7. History of esophagitis, gastritis, peptic ulcer, gastro-esophageal reflux, gastrointestinal bleeding, rectal bleeding or other clinically significant gastrointestinal abnormalities within past 3 months.
8. History of cardiovascular disease such as uncontrolled hypertension, myocardial infarction, stroke or transient ischemic attack within the past 6 months prior to screening, congestive heart failure, angina pectoris, and arrhythmia.
9. Evidence of vasospastic disease (i.e., Buerger's disease) on medical history and physical examination.
10. Unable or unwilling to abstain from methylxanthines for 72 hours pre-dose.
11. Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin, whichever is the longer) before administration of IMP in this study, at the discretion of the investigator.
12. Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
13. A major illness during the 3 months before commencement of the screening period.
14. History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
15. History of bronchial asthma or any other bronchospastic disease.
16. History of convulsions.
17. History of porphyria.
18. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
19. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
20. Diagnosis of hypotension made during the screening period.
21. Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
22. Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
23. Positive testing for HIV, Hepatitis B and Hepatitis C.
24. Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
25. Positive pregnancy test.
26. Unable or unwilling to discontinue cigarette smoking for 36 hours prior to IMP administration until 24 hours after administration of IMP of each treatment period.
27. Presence of oral or pharyngeal ulceration, inflammation or other oral pharyngeal diseases.
28. History of clinically significant autoimmune, dermatological, hematological, metabolic, neurological, psychiatric, or pulmonary disorders at discretion of the investigator.
29. Are presently using buproprion (Wellbutrin® or Zyban®), varenicline (Chantix®), xanthine-derived bronchodilators (e.g., theophylline), sympathomimetic agents, or alpha-adrenergic blocking agents.
30. Have used narcotics, antidepressants, or anxiolytics within 30 days of first receiving the IMP.
31. Presence of gum disease, temporomandibular joint dysfunction, or xerostomia.
32. Presence of tongue piercings or other foreign objects likely to interfere with dissolution procedure of IMP in the opinion of the investigator.
33. Use of St. John's Wort or kava-kava within 3 months prior to screening.
34. History of malignancy including leukemia and lymphoma (except basal cell skin cancer) within the past 5 years prior to screening.
35. Vegetarian or any abnormal diet (for whatever reason).
36. Any condition not identified in the protocol that in the opinion of the investigator or the sponsor would confound the evaluation and interpretation of the study data.
37. Any specific investigational product safety concern.
38. Vulnerable subjects, e.g., persons in detention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Maximum observed plasma concentration (Cmax)
AUC0-t | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Area under the plasma concentration versus time curve, from time zero to t, where t is the time of the last quantifiable concentration (AUC0-t)

SECONDARY OUTCOMES:
Tmax | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Time to maximum observed plasma concentration (tmax)
AUC0-inf | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Area under the plasma concentration versus time curve, with extrapolation to infinity (AUC0-inf)
λz | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Terminal elimination rate constant (λz)
t½.z | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Apparent terminal elimination half-life (t½.z)
kel | Blood samples taken pre-dose and post-dose at 5, 10, 20, 30, 40, and 50 minutes, and 1, 1.25, 1.5, 2, 3, 6, 9, 12, 16 and 24 hours
  Apparent terminal elimination rate constant (kel)

CONTACTS AND LOCATIONS:
Overall Officials: Yolandi Swart, Dr., Principal Investigator — PAREXEL (South Africa)
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, South Africa